CLINICAL TRIAL: NCT01780532
Title: Pilot Photoacoustic Imaging (PAI) of Suspicious Breast Cancers - A Clinical Feasibility Study
Brief Title: Photoacoustic Imaging (PAI) of Suspicious Breast Cancers - A Clinical Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanjiv Sam Gambhir, Chair, Dept. of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRS0018; SU-09022011-8372 (Other: Stanford University); 21623 (Other: Stanford IRB)
Record Dates: First submitted 2011-11-14; First posted 2013-01-31 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photo Acoustic Imaging (Experimental): An exploratory, single armed, pilot study designed to evaluate the feasibility of Photo Acoustic Imaging (PAI) in a clinical setting.
  Interventions: Procedure: Photoacoustic Imaging (PAI)

INTERVENTIONS:
Procedure: Photoacoustic Imaging (PAI) — Standard of Care
  Other Names: Hand held photoacoustic probe

SUMMARY:
After locating the suspicious lesion/mass with standard of care mammography and/or ultrasound, a photoacoustic scan will be performed in the breast where the lesion is located. After the PA scan a biopsy will be performed, if clinically indicated (based on the mammogram and ultrasound only).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a breast lesion/mass found at physical examination, mammography or ultrasound (US), that has not been surgically resected
* Patients may have any of the following characteristics:

  * Taking hormones (e.g., contraceptives, hormone replacement therapy, post-cancer Tamoxifen)
  * Breast implants
  * Previous breast biopsy
  * Previous breast surgery
  * Previous breast cancer
  * High risk of breast cancer (e.g., breast cancer susceptibility gene (BRCA) mutations, other gynecologic cancer)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had primary surgical excision of the suspicious finding
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The lesion visibility on PAI, described using a five-level scale: 1. Not visible 2. Barely visible 3. Fair (or moderately visible) 4. Visible 5. Clearly visible. | 6 months

SECONDARY OUTCOMES:
Measures of hypoxia in the lesion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Gambhir, MD, Principal Investigator — Stanford University